CLINICAL TRIAL: NCT02045667
Title: Combining N-of-1 Trials to Estimate Population Clinical and Cost-effectiveness of Drugs Using Bayesian Hierarchical Modeling. The Case of Mexiletine for Patients With Non- Dystrophic Myotonia.
Brief Title: Combined N-of-1 Trials Mexiletine vs Placebo in Patients With Non-Dystrophic Myotonia (NDM)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: ZonMw: The Netherlands Organisation for Health Research and Development (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Mexiletine20142015; 2010-024026-38 (EudraCT Number)
Record Dates: First submitted 2013-11-18; First posted 2014-01-27 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2016-01

CONDITIONS: Non Dystrophic Myotonia
Keywords: Becker's myotonia congenita (BMC); Thomson's myotonia congenita (TMC); Paramyotonia Congenita (PMC); Sodium Channel Myotonia (SCM)
MeSH Terms: conditions — Myotonic Disorders; Potassium aggravated myotonia | interventions — Mexiletine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): Placebo tablets three times daily orally
  Interventions: Drug: Mexiletine; Drug: Placebo
- Mexiletine (Active Comparator): Mexiletine 200mg three times daily orally
  Interventions: Drug: Mexiletine; Drug: Placebo

INTERVENTIONS:
Drug: Mexiletine — Mexiletine is a lidocaine-derivate and belongs to the class of 1B antiarrhythmic agents (Vaughan-Williams Classification of Antiarrhytmica). Class I antiarrhythmics have membrane-stabilizing properties. Drugs in this class work by interfering with the fast influx of sodium by inhibition of sodium ionchannels during the fast depolarization phase, thereby decreasing the maximal voltage and upshoot phase of the action potential.
  Mexiletine study-medication will be purchased from Stabilimento Chimico Farmaceutico Militare, Firenze, Italy.
  Other Names: Mexitil; Ritalmex
Drug: Placebo — Placebo tablets do not contain any active medicinal component.
  Other Names: Dummy; Control-arm medication

SUMMARY:
The main objective of this study is to explore whether multiple trials with individual patients (N-of-1 trials) can produce a reliable evidence base for coverage decisions on clinical and cost-effectiveness of drug treatment for patients with rare diseases. As a case study, we will study the clinical and cost-effectiveness of Mexiletine in patients with Non-Dystrophic myotonia. The results of this analysis will be compared with the results obtained from a recently published international, multi-centre, randomized, placebo-controlled trial of Mexiletine in patients with Non-Dystrophic Myotonia (clinicaltrials.gov Identifier: NCT00832000).

The secondary objective of this proposal is to assess whether mexiletine improves myotonia measured (both quantitatively and qualitative) in patients with non-dystrophic myotonia.

DETAILED DESCRIPTION:
Rationale: A current problem in the context of a coverage decision for the use of mexiletine for NDM patients is the lack of a sufficient evidence base. An innovative trial design could facilitate in establishing such an evidence base in a small group of rather heterogeneous patients. As more than 7000 rare diseases in Europe and the USA suffer from a similar lack of treatment evidence, more experience with this innovative trial design would be very helpful.

Study design: A double-blind, randomized and placebo-controlled combined N-of-1- trial using a Bayesian statistical approach.

Study population: Non-dystrophic myotonia (NDM) patients, at least 18 years old, with a genetically confirmed diagnosis.

Intervention: Each N-of-1 trial consists out of a minimum of one, and a maximum of 4 treatment sets, each comprising a 4-week period of active treatment (Mexiletine) and a 4-week period of treatment with placebo, in random order, with one week for wash-out in between. Within each mexiletine period, treatment dosage of mexiletine will be built up from 200 mg 1 time a day PO on the first day of the first week, to 200 mg 2 times a day on the second day of the first week, to the desired dosage of 200 mg 3 times a day PO on the third day of the first week and throughout the remaining days of the 4-week treatment period. A similar build-up scheme will be used within each placebo period.

Main study parameters/endpoints: The primary outcome measure for this study is a decrease in the most prominent clinical symptom: stiffness. Stiffness will be quantified by an Interactive Voice Response System (IVR) in which the patient will rate their mean daily IVR participant-assessed severity of stiffness on an ordinal scale (1-9). The secondary outcome measures will include changes in pain, weakness, and fatigue on IVR, Individual Neuromuscular Quality of Life (INQoL), the Short Form (36) Health Survey (SF-36) a patient-reported survey of patient health, blood plasma levels of mexiletine, clinical myotonia assessments, quantitative handgrip myotonia, biceps force test and needle-electromyography (EMG).

Nature and extent of the burden and risks associated with participation, benefit and group relatedness: In the screening phase, electrocardiography (ECG) and EMG recordings, laboratory values and baseline blood plasma levels of mexiletine will be tested. Medical history and written consent will also be obtained in this phase. Patients will be asked to visit the department of Neurology between 4-16 visits (depending on number of treatment sets necessary to obtain enough evidence) during the study enrolment. Each visit will approximately cost 2 hours; within each visit two questionnaires (INQoL, SF-36) need to be filled, blood plasma levels of mexiletine will be measured and clinical and electrophysiological myotonia tests need to be performed. Furthermore, an ECG and EMG will be recorded at the end of each treatment or placebo period. In addition, patients will have to call in to an interactive voice response system to report their mean daily IVR participant-assessed severity of stiffness once a week in every first and second week and daily in every third and fourth week of each treatment or placebo period.

ELIGIBILITY:
Inclusion Criteria:

1. At least 18 years of age
2. Genetically confirmed diagnosis of NDMs
3. Participation in the "Genetical variability of the Non-dystrophic Myotonia" study of J. Trip or a new patient with genetically confirmed NDM.

Exclusion Criteria:

1. Inability or unwillingness to provide informed consent.
2. Other neurological conditions that might affect the assessment of the study measurements.
3. Genetic confirmed Myotonic Dystrophy type 1 (DM1) (CTG > 50 repeats), or Myotonic Dystrophy type 2 (DM2).
4. Patients with existing cardiac conduction defects, evidenced on ECG including but not limited to the following conditions: malignant arrhythmia or cardiac conduction disturbances (such as second degree AV block, third degree atrio-ventricular (AV) block, or prolonged QT interval >500 ms or QRS duration > 150 msec).
5. Current use of the following antiarrhythmic medication for a cardiac disorder:flecainide acetate, encainide, disopyramide, procainamide, quinidine, propafenone or mexiletine.
6. Women who are pregnant or lactating.
7. Patients currently on medications for myotonia such as phenytoin and flecainide acetate within 5 days of enrollment, carbamazepine and mexiletine within 3 days of enrollment, or propafenone, procainamide, disopyramide, quinidine and encainide within 2 days of enrollment.
8. Patients with renal or hepatic disease, heart failure, history of myocardial infarction, or seizure disorders.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2014-01; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Change in patient-reported Stiffness on the IVR | Weeks 3-4 of each period - up to 44 weeks.
  Stiffness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of stiffness for each participant will be calculated form daily calls made in weeks 3-4 of each period.

SECONDARY OUTCOMES:
Change in Individualized Neuromuscular Quality of Life Scale - Summary Score | Week 4 of each period - up to 44 weeks.
  Quality of life scale for patinets with neuromuscular disorders. The INQoL summary score is a weighted average made up of 5 subdomains (activities, social relationships, independence, emotions, and body image) which document the impact of a disease on a patients' quality of life. Scores range from 0-100, and can be interpreted as the percent of maximal detrimental impact on quality of life. A higher score indicates more detrimental impact.
Change in Short Form 36 - Physical Composite Score | Week 4 of each period - up to 44 weeks.
  The SF-36 is a standard quality of life instrument. The physical composite score represents the the physical burden on quality of life and is a summary of questions related to physical impact of a disease or condition (physical function, role physical, bodily pain, and general health). The score is nomralized to the population and ranges from 0-100, with the US normal value of 50. A lower score represents a greater impact of quality of life.
Change in Clinical myotonia bedside-tests (Seconds) | Week 4 of each period - up to 44 weeks.
  1. Eye closure myotonia. The participant will be instructed to close the eyes tightly for three seconds and then to open the eyes. Eye closure myotonia is present if there is difficulty fully opening the eyelids. This will be repeated for a total of 5 times. Each attempt will be timed.
  2. Hand-grip myotonia. The participant will be instructed to forcefully close the fingers in a fist for three seconds and then rapidly open the fist and extend the fingers. Hand-grip myotonia is present if the fingers cannot be immediately extended. The time it takes (in seconds) for the fingers to be fully extended will be recorded. This will be repeated for a total of 5 times. Each attempt will be timed.
  3. Percussion myotonia.
Change in Muscle relaxation times measured with quantitative grip myometry (Seconds) | Week 4 of each period - up to 44 weeks.
  Maximum Voluntary Isometric Contractions (MVIC's) of the long finger flexors and the subsequent relaxation time (myotonia) will be measured using a technique developed at the University of Rochester. To measure the extent of grip myotonia of resting forearm muscle, each participant will squeeze the grip handle with a maximum grip for 3 seconds then relax until the force returns to baseline. The time required for relaxation (the relaxation time (RT)) following this initial MVIC will be used to calculate the degree of myotonia. To determine if repeated muscle contractions shorten the time required for full muscle relaxation, eg., warm-up, a series of five MVICs will be made, each for three seconds duration followed by a ten second period of rest. The measurement of warm-up will be made by comparing relaxation time for the initial MVIC compared to the relaxation time following the final contraction in the series of five contractions used as warm-up exercise.
Change in Graded Myotonia by Needle Electromyography | Week 4 of each period - up to 44 weeks.
  Concentric needle EMG will be performed in the rectus femoris muscles. These muscle were chosen based on the data from the NDM natural history study as performed in Jeroen Trip his PhD-thesis, and will be consistent throughout this study. According to established criteria myotonic discharges will be defined and quantified: Myotonic discharges must be at least 500 msec and elicited in three areas of the muscle outside of the endplate zone. Grading of myotonic discharges: 1+: fulfills minimal requirements; 2+: myotonic discharges in more than ½ of needle locations; 3+: myotonic discharges with each needle movement in all examined areas.
Change in Mexiletine serum plasma concentration levels | Weeks 1 and 4 of each period - up to 44 weeks.
  Mexiletine serum plasma concentration levels will be measured using a High-performance liquid chromatography-technique to analyse if they are within therapeutic range and to exclude any carry-over effects.
Change in Patient-reported Pain on the IVR | Weeks 3-4 of each period - up to 44 weeks.
  Pain measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of pain for each participant will be calculated form daily calls made in weeks 3-4 of each period.
Change in Patient-reported Weakness on the IVR | Weeks 3-4 of each period - up to 44 weeks.
  Weakness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of weakness for each participant will be calculated form daily calls made in weeks 3-4 of each period.
Change in Patient-reported Tiredness on the IVR | Weeks 3-4 of each period - up to 44 weeks.
  Tiredness measured on a 1-9 scale, 1 being minimal, 9 the worst ever experienced. 0=no symptom reported. For analysis the average severity of tiredness for each participant will be calculated form daily calls made in weeks 3-4 of each period.
Change in Short Form 36 - Mental Composite Score | Week 4 of each period - up to 44 weeks.
  The SF-36 is a standard quality of life instrument. The mental composite score represents the the mental burden on quality of life and is a summary of questions related to mental impact of a disease or condition (mental function, role emotional, vitality, and mental health). The score is nomralized to the population and ranges from 0-100, with the US normal value of 50. A lower score represents a greater impact of quality of life.

OTHER OUTCOMES:
Change in ECG conduction times: PR, QRS and QTc-time | Week 4 of each period - up to 44 weeks.
  PR, QRS and QTc-times are segments of the ECG that in case of a change (increase or decrease) could hold a risk for cardiac arrhythmia.

CONTACTS AND LOCATIONS:
Overall Officials: Prof. dr. BGM van Engelen, MD, PhD, Principal Investigator — Department of Neurology, Radboud University Nijmegen Medical Centre, the Netherlands; Prof. dr. GJ van der Wilt, PhD, Principal Investigator — Department of Epidemiology, HTA and biostatistics, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. BC Stunnenberg, MD, Study Chair — Department of Neurology, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. W Woertman, PhD, Study Chair — Department of Epidemiologie, HTA and biostatistics, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. B Schouwenberg, MD, Study Chair — Department of Pharmacology and Toxicology, Radboud University Nijmegen Medical Centre, the Netherlands; Dr. G Drost, MD, PhD, Study Chair — Department of Neurology, University Medical Centre Groningen, the Netherlands; Drs. J Raaphorst, MD, Study Chair — Department of Neurology, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. N van Alfen, MD, PhD, Study Chair — Department of Neurology, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. J Timmermans, MD, Study Chair — Department of Cardiology, Radboud University Nijmegen Medical Centre, the Netherlands; Drs. H Groenewoud, MSc, Study Chair — Department of Epidemiologie, HTA and biostatistics, Radboud University Nijmegen Medical Centre, the Netherlands
Locations (1):
- Departments of Neurology, Radboud University Nijmegen Medical Centre, the Netherlands, Nijmegen, Gelderland, Netherlands

REFERENCES:
- [Derived] Stunnenberg BC, Raaphorst J, Groenewoud HM, Statland JM, Griggs RC, Woertman W, Stegeman DF, Timmermans J, Trivedi J, Matthews E, Saris CGJ, Schouwenberg BJ, Drost G, van Engelen BGM, van der Wilt GJ. Effect of Mexiletine on Muscle Stiffness in Patients With Nondystrophic Myotonia Evaluated Using Aggregated N-of-1 Trials. JAMA. 2018 Dec 11;320(22):2344-2353. doi: 10.1001/jama.2018.18020. PMID 30535218
- [Derived] Stunnenberg BC, Woertman W, Raaphorst J, Statland JM, Griggs RC, Timmermans J, Saris CG, Schouwenberg BJ, Groenewoud HM, Stegeman DF, van Engelen BG, Drost G, van der Wilt GJ. Combined N-of-1 trials to investigate mexiletine in non-dystrophic myotonia using a Bayesian approach; study rationale and protocol. BMC Neurol. 2015 Mar 25;15:43. doi: 10.1186/s12883-015-0294-4. PMID 25880166